CLINICAL TRIAL: NCT06107868
Title: Phase I Study of the PKMYT1 Inhibitor RP-6306 in Combination With Carboplatin and Paclitaxel for the Treatment of Recurrent TP53 Ovarian and Uterine Cancer
Brief Title: Phase 1 Study of RP-6306 With Carboplatin and Paclitaxel in TP53 Ovarian and Uterine Cancer
Acronym: GyneRep
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OZUHN-019; CAPCR 23-5475 (Other: University Health Network)
Record Dates: First submitted 2023-10-25; First posted 2023-10-30 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Ovarian Cancer; Recurrent Uterine Cancer; Metastatic Cancer; Advanced Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Uterine Neoplasms; Neoplasm Metastasis | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A - Dose Escalation (Experimental): RP6306, 40 mg orally, twice a day, continuously or on Days 1 to 3, for 1 or 2 weeks, every 21-day cycle.
  Carboplatin, AUC 5 intravenously, on Day 1 of every 21-day cycle.
  Paclitaxel, 175 mg/m2 intravenously, on Day 1 of every 21-day cycle.
  Interventions: Drug: RP-6306; Drug: Carboplatin; Drug: Paclitaxel
- Part B - Dose Expansion (Experimental): RP6306, 40 mg orally at the best schedule determined in Part A.
  Carboplatin, AUC 5 intravenously, on Day 1 of every 21-day cycle.
  Paclitaxel, 175 mg/m2 intravenously, on Day 1 every 21-day cycle.
  Interventions: Drug: RP-6306; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: RP-6306 — RP-6306 is a selective inhibitor of PKMYT1 kinase. RP-6306 is an investigational agent.
Drug: Carboplatin — Carboplatin is an antineoplastic agent.
Drug: Paclitaxel — Paclitaxel is an antineoplastic agent.

SUMMARY:
This is a phase 1 study to evaluate investigational drug RP-6306 in combination with carboplatin and paclitaxel in patients with TP53 mutated ovarian or uterine cancer. The dose escalation part of the study will determine the maximum tolerated dose (MTD) and recommended Phase 2 Dose (RP2D) and schedule of RP-6306 in combination with carboplatin and paclitaxel and the dose expansion will further assess the safety and tolerability as well as determine the preliminary efficacy of RP-6306 in combination with carboplatin and paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Females ≥18 years old at the time of signature of the consent form.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 28 days prior to enrollment.
* All patients must have histologically proven, locally advanced or metastatic recurrent ovarian and uterine cancer. Patients will be eligible only if available curative therapy does not exist.
* Ovarian and uterine cancer should be high-grade and TP53 abnormal by immunohistochemistry or TP53 mutated by genomic profiling.
* Patients must be eligible for re-challenge carboplatin and paclitaxel.
* Patient must have archival tissue available for molecular profiling.
* Measurable disease as per Response Evaluation Criteria in Solid Tumours (RECIST) v1.1 at the time of enrollment.
* Ability to comply with the protocol and study procedures.
* Acceptable study required organ function at screening
* Acceptable study required hematologic function at screening
* Negative pregnancy test (serum) for women of child-bearing potential (WOCBP) at screening. WOCBP who are sexually active and their partners must agree to use a highly effective form of contraception throughout their participation during the study and for 6 months after the last dose of study treatment.
* Resolution of all toxicities of prior therapy or surgical procedures to baseline or Grade 1 (except for neuropathy, hypothyroidism requiring medication, and alopecia, which must have resolved to Grade ≤2).
* Any prior radiation must have been completed at least 7 days prior to the start of study treatment, and patients must have recovered from any acute adverse effects prior to the start of study treatment.
* Life expectancy ≥12 weeks after the start of the treatment according to the Investigator's judgment.

Exclusion Criteria:

* Chemotherapy or small molecule antineoplastic agent given within 21 days or <5 half-lives, whichever is shorter, prior to first dose of study treatment.
* History or current condition (such as transfusion-dependent anemia or thrombocytopenia), or laboratory abnormality that might confound the study results, or interfere with the patient's participation for the full duration of the study treatment.
* Patients who are pregnant or breastfeeding.
* Known sensitivity to any of the ingredients of RP-6306, carboplatin and paclitaxel. Patients are eligible if pre-medications with steroids previously controlled sensitivity and patient was able to receive treatment.
* Patients who are unable to swallow oral medications.
* Prior treatment with a WEE1 inhibitor or PKMYT1 inhibitor.
* Life-threatening illness, medical condition, active uncontrolled infection, or organ system dysfunction (such as ascites, coagulopathy, or encephalopathy), or other reasons which, in the Investigator's opinion, could compromise the participating patient's safety, or interfere with or compromise the integrity of the study outcomes.
* Major surgery within 4 weeks prior to first dose of study treatment.
* Uncontrolled, symptomatic brain metastases. Patients with previously treated brain metastases may participate provided the metastases are stable, they have no evidence of new or enlarged brain metastases, and they are clinically stable and off steroids for at least 7 days prior to study treatment.
* Uncontrolled hypertension despite adequate treatment prior to first dose of study treatment.
* Gastrointestinal disorders that may significantly interfere with absorption of the study medication by Investigator's assessment.
* Active, uncontrolled bacterial, fungal, or viral infection, including hepatitis B virus, hepatitis C virus, known human immunodeficiency virus (HIV), or AIDS-related illness. In equivocal cases, patients whose viral load is negative may be eligible. HIV seropositive patients who are healthy and low risk for AIDS-related outcomes could be considered eligible.
* Moderate or severe hepatic impairment (ie, Child-Pugh Class B or C) at the time of registration.
* Any of the following cardiac diseases currently or within the last 6 months as defined by New York Heart Association (NYHA) ≥Class 2:

  1. Unstable angina pectoris
  2. Congestive heart failure
  3. Acute myocardial infarction
  4. Conduction abnormality not controlled with pacemaker or medication
  5. Significant ventricular or supraventricular arrhythmias (patients with chronic rate-controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible)
  6. Clinically relevant electrolyte abnormalities
* Current treatment with medications that are well-known to prolong the QT interval.
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol and/or follow-up procedures outlined in the protocol.
* Patients who are receiving strong CYP3A inhibitors or inducers within 14 days prior to first dose of study treatment, investigational therapy or anticancer agents, or antiviral therapies that are sensitive CYP3A substrates.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of dose-limiting toxicities (DLTs) at Dose Level 1 | 21 days
Frequency of dose-limiting toxicities (DLTs) at Dose Level 2 | 21 days
Frequency of dose-limiting toxicities (DLTs) at Dose Level -1 | 21 days
Frequency of dose-limiting toxicities (DLTs) at Dose Level -2 | 21 days

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | 4 years
Progression-free survival | 6 months
  Time from the first day of study treatment to disease progression.
Objective response rate | 4 years
  Proportion of patients with confirmed complete response (CR) or partial response (PR)
Disease Control Rate | At least 4 months after first dose of study treatment
  Proportion of patients with a confirmed best response of CR or PR, or stable disease
Duration of Response | 4 years
  Time interval between the date of the earliest qualifying response (CR or PR) and the date of disease progression or death for any cause, whichever occurs earlier
Average change in tumour size | 4 years
Plasma concentrations of RP-6306 | Cmax, time to Tmax

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Lheureux, MD, Principal Investigator — The Princess Margaret Cancer Foundation
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No